CLINICAL TRIAL: NCT00251290
Title: Diagnosis and Treatment of Sleep-Disordered Breathing in the Homes of Patients With Transient Ischemic Attack
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Robert Wood Johnson Foundation (Other); ResMed Foundation (Other); US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Dawn M. Bravata, M.D., Roudebush VAMC
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RWJ-GPFS-051081
Record Dates: First submitted 2005-11-07; First posted 2005-11-09 (Estimated); Last update posted 2009-03-03 (Estimated); Status verified 2009-03

CONDITIONS: Transient Ischemic Attack; Sleep Apnea
Keywords: transient ischemic attack; sleep apnea
MeSH Terms: conditions — Ischemic Attack, Transient; Sleep Apnea Syndromes

INTERVENTIONS:
Procedure: auto-titrating continuous positive airway pressure — Continuous positive Airway pressure (CPAP) use for 90 days post TIA

SUMMARY:
Generalist physicians in the outpatient setting care for 80% of the 300,000 patients who have transient ischemic attacks (TIA) annually in the United States. Despite existing secondary prevention therapies, recurrent ischemic events are common following a TIA. Given the risk of poor outcomes and the important role of the generalist, new therapeutic approaches for patients with TIA are needed that can be applied by generalists to outpatients. This research will develop and evaluate a new therapeutic approach that centers on the observations that sleep-disordered breathing is a risk factor for cerebrovascular and cardiovascular disease, is common in patients with cerebrovascular disease, and is associated with poor outcome following a stroke or TIA. We posit that diagnosing and treating sleep-disordered breathing in the home of TIA patients can improve cerebrovascular and cardiovascular outcomes.

The primary aims are to determine in TIA patients: 1) the prevalence of sleep-disordered breathing, 2) the feasibility of diagnosing and treating sleep-disordered breathing using an auto-titrating continuous positive airways pressure (auto-CPAP) machine within 24-hours of TIA symptom onset, 3) adherence to auto-CPAP, and 4) the effect of auto-CPAP on blood pressure.

We will recruit 80 TIA patients to be randomly assigned to either the intervention or the control groups. Each patient in the intervention group will use an auto-CPAP machine for up to 90 days and will then receive an unattended sleep study using a sleep monitor. Each patient in the control group will receive two unattended sleep studies, one upon enrollment and another after 90 days.

ELIGIBILITY:
Inclusion Criteria: transient ischemic attack - Exclusion Criteria:age <45 years; respiratory distress or known sleep-disordered breathing; chronic obstructive pulmonary disease (COPD) requiring oxygen; pregnancy; time from symptom onset to beginning of study intervention 72 hours; life expectancy <6 months; cognitive impairment (Mini-Mental Status Exam<20); inability to provide informed consent; inability to communicate in English; residence outside the greater New Haven area; or any condition where the monitoring required by the study would constitute a risk to the patient or impair his or her care.

-

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2004-11; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
prevalence of sleep-disordered breathing in patients with TIA, proportion of patients who use auto-CPAP >4 hours per night, and change in systolic blood pressure | 90 days

SECONDARY OUTCOMES:
Recurrent vascular events (transient ischemic attack, stroke, myocardial infarction, congestive heart failure requiring hospitalization, and death), sleepiness, cognition, depression, functional status, and quality of life. | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Dawn M Bravata, MD, Principal Investigator — Yale School of Medicine; VA Connecticut Healthcare System
Locations (3):
- United States (3):
  - Hospital of St. Raphael, New Haven, Connecticut
  - Yale-New Haven Hospital, New Haven, Connecticut
  - VA Connecticut Healthcare System, West Haven Campus, West Haven, Connecticut